CLINICAL TRIAL: NCT00021333
Title: Phase II Evaluation Of Paclitaxel And Cisplatin In Combination With Split Course Hyperfractionated Radiation Therapy And Granulocyte-Colony Stimulating Factor In Previously Irradiated Patients With Locally Recurrent Carcinoma Of The Head And Neck, And Lung
Brief Title: Paclitaxel and Cisplatin Plus Radiation Therapy Followed by Filgrastim in Treating Patients With Recurrent Head and Neck Cancer or Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068770; P30CA006927 (NIH); FCCC-99025; NCI-G01-1983
Record Dates: First submitted 2001-07-11; First posted 2004-01-14 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: recurrent non-small cell lung cancer; recurrent small cell lung cancer; recurrent thyroid cancer; recurrent salivary gland cancer; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thyroid Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — Filgrastim; Cisplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may make tumor cells more sensitive to radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel and cisplatin plus radiation therapy followed by filgrastim in treating patients who have recurrent head and neck cancer or lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with locally recurrent carcinoma of the head and neck or lung treated with paclitaxel and cisplatin with concurrent radiotherapy followed by filgrastim (G-CSF). II. Assess the toxicity of this regimen in these patients. III. Determine the time to progression and the sites and pattern of progression in patients treated with this regimen. IV. Determine the median, 1-year, and 2-year survival rates of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (squamous cell carcinoma of the head and neck vs salivary gland malignancy or other non-squamous cell carcinoma of the head and neck vs lung cancer). Patients receive paclitaxel IV over 1 hour and cisplatin IV over 30-120 minutes on days 1-5. Patients undergo radiotherapy twice daily on days 1-5. Patients receive filgrastim (G-CSF) subcutaneously on days 6-13 or until blood counts recover. Treatment repeats every 2 weeks for a total of 4 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 42-84 patients (14-28 per stratum) will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of 1 of the following: Previously irradiated, locally recurrent squamous cell carcinoma of the head and neck (SCCHN) or head and neck skin/appendages with no distant metastases New second or subsequent primary SCCHN in a previously irradiated field with no distant metastases Salivary gland malignancy or other non-squamous cell primary head and neck cancer Previously irradiated, locally recurrent carcinoma of the lung No clinical evidence of symptomatic bone or brain metastases requiring radiotherapy No leptomeningeal metastases requiring intrathecal therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No active, uncontrolled congestive heart failure or arrhythmia within the past 6 months Other: No pre-existing neuropathy grade 2 or greater interfering with daily activities No prior allergy to drugs using Cremophor EL No hypersensitivity to E. coli-derived proteins No significant concurrent medical or psychiatric disorder that would preclude study No other condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 months since prior radiotherapy Prior or concurrent cumulative radiotherapy dose to spinal cord no greater than 5,000 cGy Surgery: Not specified Other: Concurrent beta-blockers, digitalis derivatives, or calcium-channel blocking agents allowed if cardiac conditions are stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1999-09; Primary Completion 2006-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (18):
- United States (18):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - Central Montgomery Medical Center, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Southern Chester County Medical Center, West Grove, Pennsylvania